CLINICAL TRIAL: NCT02026635
Title: Cardiac Compass With Optivol® to Negate Future Inpatient Re-admissions Through Monitoring in Heart Failure Patients (CONFIRM-HF)
Brief Title: Cardiac Compass With Optivol® to Negate Future Inpatient Re-admissions Through Monitoring in HF Patients (CONFIRM-HF)
Acronym: CONFIRM-HF
Status: Withdrawn | Type: Observational
Why Stopped: No subjects enrolled
Sponsor: Thomas Jefferson University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 13P.296
Record Dates: First submitted 2013-12-16; First posted 2014-01-03 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Heart Failure
Keywords: heart failure; Optivol® cardiac device; Medtronic CareLink
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Optivol® Device in CareLink: A single cohort group of heart failure patients with already implanted Optivol® capable devices who are discharged home from the hospital

SUMMARY:
A research study to determine if heart failure can be medically managed using data collected from cardiac monitoring devices

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Admission for worsening of HF
* Discharged to home
* Have appropriate cardiac device with OptiVol® implanted for at least 34 days prior to enrollment
* Enrolled in Carelink® system and able to transmit data
* Able to participate for at least 3 months

Exclusion Criteria:

* Post heart transplant or actively listed
* End-stage (Stage D) HF, including treatment with chronic ionotropic drugs or left ventricular assist device support
* Stage IV or V chronic renal dysfunction (GFR <25 mol/min per 1.73 M2)
* Severe Chronic Obstructive Pulmonary Disease (COPD) requiring home oxygen
* Severe pulmonary hypertension not due to left-sided HF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital inpatients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Physician Use of Cardiac Compass Reports to Determine HF Treatment Decisions | 90 days from enrollment
  Assessment will be completed at time of enrollment and days 3 to 7, 14 to 21, 30 and 90 post discharge.

SECONDARY OUTCOMES:
Heart Failure Clinical Events | 90 days from enrollment
  Track HF re-admissions and other clinical encounters between 30 and 90 days post discharge for HF.
Assess Patient-Reported Quality of Life | 90 days from enrollment
  Assess the association between the use of Cardiac Compass Report and OptiVol® and improved HF patient quality of life at both time points (30 and 90 days post discharge) utilizing the Kansas City Cardiomyopathy Questionnaire (KCCQ)

CONTACTS AND LOCATIONS:
Overall Officials: David J Whellan, MD MHS, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States